CLINICAL TRIAL: NCT03680885
Title: Reliability Testing of a Non-invasive, Pain-free, Taste-based Assessment Approach to Lidocaine Effectiveness
Brief Title: Validating a New Non-invasive Approach to Testing Lidocaine Effectiveness
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: PhenoSolve, LLC (Industry)
Collaborators: Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2018-271
Record Dates: First submitted 2018-09-17; First posted 2018-09-21 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: ADHD; Controls
Keywords: Lidocaine ineffectiveness; ADHD; ADD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Half the subjects will have a self-reported history of lidocaine working for them (effective) and half will have a history of difficulty getting numb (ineffective).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The scoring of the lidocaine test is masked, using the coded identity of the tastes. The tastes will be assessed in random order. Each subject will have 2 tests with lidocaine gel and 2 with a placebo gel, in random order, each on different days. The subjects and other study personnel will be told not to discuss what the subject could or couldn't taste. Scoring will be done only after all testing on the subject is complete. A person not involved in the testing will keep track of which gels the subject has had.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Reports getting numb at dentist (Active Comparator): Subjects will be tested twice with lidocaine gel, twice with a Placebo and once with Injected Lidocaine to assess effectiveness of lidocaine. Each assessment will be on a different day.
  Interventions: Drug: Lidocaine gel; Drug: Placebo; Drug: Injected lidocaine
- Reports trouble getting numb at dentist (Active Comparator): Subjects will be tested twice with lidocaine gel, twice with a Placebo and once with Injected Lidocaine to assess effectiveness of lidocaine. Each assessment will be on a different day.
  Interventions: Drug: Lidocaine gel; Drug: Placebo; Drug: Injected lidocaine

INTERVENTIONS:
Drug: Lidocaine gel — Lidocaine gel 5%, PEG with FD&C Blue No.1 (Brilliant Blue FCF)
  Other Names: Intervention
Drug: Placebo — PEG with FD&C Blue No.1 (Brilliant Blue FCF)
  Other Names: Control gel
Drug: Injected lidocaine — Standard FDA-approved dental injectable lidocaine
  Other Names: Current practice

SUMMARY:
This work will assess the reliability of a simple painless test for the effectiveness of the commonly used local anesthetic lidocaine

DETAILED DESCRIPTION:
In prior tests with a convenience sample, subjects who reported that they had no trouble getting numb at the dentist, also got numb with lidocaine gel on the surface of the tongue. That numbness prevented them from being able to taste any flavor until the numbness had worn off. Subjects who reported having trouble getting numb at the dentist, could still taste flavors after the application of lidocaine.

This work will assess the reliability of a taste-based approach for creating a non-invasive way to test lidocaine effectiveness. The controlled trial will assess the ability of lidocaine oral gel to block taste (e.g., sweet) in 20 adults (ages 18-49) half with history of trouble getting numb at the dentist (Arm 2) and half with no trouble (Arm 1). To determine reproducibility, the taste-based test will be done 4 times on different days, twice with lidocaine and twice with a placebo, with randomization and double-blinding. These repeated results will be compared to a fifth assessment, against the "gold standard" of injection of lidocaine, assessed using a dental probe.

On each of four separate visits, in randomized order, the subject will be tested with tastants to the tongue twice after application of a lidocaine gel to the tongue and twice with a placebo gel. After a wait of two-minutes, the three tastants will be tested. The subject is blinded to the taste and the identity of the gel, which have been compounded to look the same.

On the fifth (last) visit, the subject will get an oral injection of lidocaine and the numbness assessed.

The results across the five tests will then be analyzed.

We are testing in separate studies NCT 03563573 and NCT 03676725 the prevalence of lidocaine ineffectiveness in those with Attention Deficit Hyperactivity Disorder (ADHD) and in the general population without ADHD. We believe the prevalence will be higher in ADHD. As a result, in this evaluation we have one Arm "gets numb at the dentist" where exclusion criteria includes ADHD and a second Arm "has trouble getting numb at the dentist" that does not have that exclusion.

ELIGIBILITY:
Arm 1 Eligibility

Inclusion Criteria:

- Report "get numb at dentist"

Exclusion Criteria:

* ADHD, ADD, and other inattention disorders
* Known adverse reactions to lidocaine;
* Epilepsy
* IQ <80
* Severe head trauma
* Birth weight <2270 grams
* Severe autism
* Generalized anxiety disorders (but dental-specific anxiety will not be an exclusion because many of these individuals may be ones with anxiety because of painful dental experiences with lidocaine ineffectiveness)
* Mouth sores
* Ehlers Danlos syndrome
* Red hair
* Current pregnancy
* Treatment currently with potassium or potassium-elevating drugs such as renin-angiotensin-aldosterone blockers

Angiotensin Converting Enzyme Inhibitors

* Alacepril (not available in US)
* Benazepril (Lotensin)
* Captopril (trade name Capoten)
* Cilazapril (Inhibace)
* Delapril (not available in US)
* Enalapril (Vasotec/Renitec)
* Fosinopril (Fositen/Monopril)
* Imidapril (Tanatril)
* Lisinopril (Listril/Lopril/Novatec/Prinivil/Zestril)
* Moexipril (Univasc)
* Perindopril (Coversyl/Aceon/Perindo)
* Quinapril (Accupril)
* Ramipril (Altace/Prilace/Ramace/Ramiwin/Triatec/Tritace)
* Spirapril (Renormax)
* Temocapril (not available in US)
* Teprotide (but not active by oral administration and not used in US)
* Trandolapril (Mavik/Odrik/Gopten)
* Zofenopril

Angiotensin receptor blockers

* Azilsartan (Edarbi)
* Candesartan (Atacand)
* Eprosartan (Teveten)
* Fimasartan (Kanarb)
* Irbesartan (Avapro)
* Losartan (Cozaar)
* Olmesartan (Benicar/Olmetec)
* Telmisartan (Micardis)
* Valsartan (Diovan)

Aldosterone antagonists

* Spironolactone (Aldactone)
* Eplerenone (Inspra)

Renin inhibitors - Aliskiren (Tekturna, Rasilez)

Other potassium elevating agents

* Antibiotics, including penicillin G and trimethoprim
* Azole antifungals
* Beta-blockers
* Herbal supplements, including milkweed, lily of the valley, Siberian ginseng, Hawthorn berries
* Heparin
* Nonsteroidal anti-inflammatory medications (NSAIDs)
* Oral contraceptives containing drospirenone

Arm 2 Eligibility

Inclusion Criteria:

- Report "trouble getting numb at dentist"

Exclusion Criteria:

* Known adverse reactions to lidocaine;
* Epilepsy
* IQ <80
* Severe head trauma
* Birth weight <2270 grams
* Severe autism
* Generalized anxiety disorders (but dental-specific anxiety will not be an exclusion because many of these individuals may be ones with anxiety because of painful dental experiences with lidocaine ineffectiveness)
* Mouth sores
* Ehlers Danlos syndrome
* Red hair
* Current pregnancy
* Treatment currently with potassium or potassium-elevating drugs such as renin-angiotensin-aldosterone blockers

Angiotensin Converting Enzyme Inhibitors

* Alacepril (not available in US)
* Benazepril (Lotensin)
* Captopril (trade name Capoten)
* Cilazapril (Inhibace)
* Delapril (not available in US)
* Enalapril (Vasotec/Renitec)
* Fosinopril (Fositen/Monopril)
* Imidapril (Tanatril)
* Lisinopril (Listril/Lopril/Novatec/Prinivil/Zestril)
* Moexipril (Univasc)
* Perindopril (Coversyl/Aceon/Perindo)
* Quinapril (Accupril)
* Ramipril (Altace/Prilace/Ramace/Ramiwin/Triatec/Tritace)
* Spirapril (Renormax)
* Temocapril (not available in US)
* Teprotide (but not active by oral administration and not used in US)
* Trandolapril (Mavik/Odrik/Gopten)
* Zofenopril

Angiotensin receptor blockers

* Azilsartan (Edarbi)
* Candesartan (Atacand)
* Eprosartan (Teveten)
* Fimasartan (Kanarb)
* Irbesartan (Avapro)
* Losartan (Cozaar)
* Olmesartan (Benicar/Olmetec)
* Telmisartan (Micardis)
* Valsartan (Diovan)

Aldosterone antagonists

* Spironolactone (Aldactone)
* Eplerenone (Inspra)

Renin inhibitors

- Aliskiren (Tekturna, Rasilez)

Other potassium elevating agents

* Antibiotics, including penicillin G and trimethoprim
* Azole antifungals
* Beta-blockers
* Herbal supplements, including milkweed, lily of the valley, Siberian ginseng, Hawthorn berries
* Heparin
* Nonsteroidal anti-inflammatory medications (NSAIDs)
* Oral contraceptives containing drospirenone

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Taste sensation after lidocaine or placebo | 4 visits each of 30 minutes within weeks of one another, average ~1 month total
  The subject is blinded to the tastant and gel identities. The 3 tastants are tested in randomized order.
  After application of lidocaine gel or placebo to the tongue, and a wait of 2 minutes, the subject's tongue is rubbed with a swab that has been wet with the tastant on the subject's tongue.
  The subject is asked to identify the taste (e.g., sweet).
  Then, on a 5-point scale (0-4, ranging from none to very intense) they are asked to rate the intensity of the taste.
  The process is repeated for each of the three tastants.
  The consistency of the subject responses over the 4 sessions will be analyzed.
Ability to feel pressure and discomfort after injection of lidocaine into the cheek | 1 visit of 30 minutes after other 4 visits, average ~1 month total
  Inject lidocaine as would be done in a dental visit, assess numbness to pressure and discomfort using the Baker Wong FACES scale (0-10) scale of discomfort, ranging from none to intense pain.
  The effectiveness of lidocaine will be assessed, and then the results compared to Outcome 1.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Segal, MD PhD, Principal Investigator — PhenoSolve, LLC
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share with the FDA the validation of the taste approach to testing lidocaine effectiveness, as part of an IDE application.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 9-12 months

REFERENCES:
- [Result] Infante MA, Moore EM, Nguyen TT, Fourligas N, Mattson SN, Riley EP. Objective assessment of ADHD core symptoms in children with heavy prenatal alcohol exposure. Physiol Behav. 2015 Sep 1;148:45-50. doi: 10.1016/j.physbeh.2014.10.014. Epub 2014 Oct 23. PMID 25447751
- [Result] Levitt JO. Practical aspects in the management of hypokalemic periodic paralysis. J Transl Med. 2008 Apr 21;6:18. doi: 10.1186/1479-5876-6-18. PMID 18426576
- [Result] Nakai Y, Milgrom P, Mancl L, Coldwell SE, Domoto PK, Ramsay DS. Effectiveness of local anesthesia in pediatric dental practice. J Am Dent Assoc. 2000 Dec;131(12):1699-705. doi: 10.14219/jada.archive.2000.0115. PMID 11143733
- [Result] Segal MM. We cannot say whether attention deficit hyperactivity disorder exists, but we can find its molecular mechanisms. Pediatr Neurol. 2014 Jul;51(1):15-6. doi: 10.1016/j.pediatrneurol.2014.04.014. Epub 2014 Apr 18. No abstract available. PMID 24938135
- [Result] Segal MM, Rogers GF, Needleman HL, Chapman CA. Hypokalemic sensory overstimulation. J Child Neurol. 2007 Dec;22(12):1408-10. doi: 10.1177/0883073807307095. PMID 18174562
- [Result] Segal MM, Douglas AF. Late sodium channel openings underlying epileptiform activity are preferentially diminished by the anticonvulsant phenytoin. J Neurophysiol. 1997 Jun;77(6):3021-34. doi: 10.1152/jn.1997.77.6.3021. PMID 9212254
- [Result] Teicher MH, Polcari A, Fourligas N, Vitaliano G, Navalta CP. Hyperactivity persists in male and female adults with ADHD and remains a highly discriminative feature of the disorder: a case-control study. BMC Psychiatry. 2012 Nov 7;12:190. doi: 10.1186/1471-244X-12-190. PMID 23134619
- See also: Saul R (2014) "ADHD Does Not Exist". HarperCollins — https://www.amazon.com/ADHD-Does-Not-Exist-Hyperactivity/dp/006226673X
- See also: Rozanski RJ, Primosch RE, Courts FJ (1988). Clinical efficacy of 1 and 2% solutions of lidocaine. Pediatr Dent.10:287-90 — https://pdfs.semanticscholar.org/1778/f693dc7dd257ab98a96b5bf03408d9cef3eb.pdf
- See also: Segal MM, Jurkat-Rott K, Levitt J, Lehmann-Horn F (2014) Hypokalemic periodic paralysis - an owner's manual — https://www.uni-ulm.de/fileadmin/website_uni_ulm/med.inst.040/Dokumente/owner.html
- See also: Segal MM (2015) Devices, Kits, and Methods for Determining Sensitivity to Anesthetics. US Patent Filing 62/210,747, Filed 09/14/2015 — https://patents.google.com/patent/WO2017035470A1/en